CLINICAL TRIAL: NCT05474261
Title: Clinical Usefulness of the Valsalva Maneuver to Improve Hemostasis During Thyroidectomy
Brief Title: Valsalva Maneuver in Thyroidectomy
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Mario Pacilli, Principal Investigator, University of Foggia
Other Study IDs: UFoggia2
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: The Role of Valsalva Manoeuvre, in Thyroidectomy to Reduce Postoperative Bleeding
MeSH Terms: interventions — Valsalva Maneuver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP A-NO Valsalva maneuver
- GROUP B- Valsalva maneuver
  Interventions: Procedure: Valsalva maneuver

INTERVENTIONS:
Procedure: Valsalva maneuver — Valsalva maneuver: increase intrabdominal pressure
  Groups: GROUP B- Valsalva maneuver

SUMMARY:
Bleeding after total thyroidectomy remains a rare event that affects early postoperative morbidity, occurring in 0.3% up to 4.2% of cases. Intraoperative bleeding is an unpleasant complication, and it is often easily manageable though postoperative bleeding may represent a life-threatening condition for the patient.

Between January 2019 to February 2022 , 250 consecutive patients were listed for thyroidectomy. The Investigators selected 178 patients and divided them in two groups based on the execution of the Valsalva Manoeuvre.

The purpose of the investigator is to clarify whether the routine intraoperative execution of a Valsalva manoeuvre (VM) may affect the detection of bleeding that would otherwise remain occult and therefore may manifest in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* thyroid diseases

Exclusion Criteria:

* lymph node dissection
* minimally invasive approaches
* high anesthesiological risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients underwent total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Volume of cervical drainage after total thyroidectomy | 24 hours
  Bleeding after thyroidectomy is evaluated based on the total volume of cervical drainage output (ml)
Number of reinterventions | 24 hours
  Reoperations to resolve post thyroidectomy bleeding, which can cause airway compression and choking signs and symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Di Foggia, Foggia, Italy

DOCUMENTS (1):
  • Study Protocol (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT05474261/Prot_000.pdf